CLINICAL TRIAL: NCT04773054
Title: Application of Advanced High-sensitivity Technologies for Identifying Infections in Patients With Aseptic Loosening of Hip Arthroplasty.
Brief Title: Identification of Infections in Hip Arthroplasty Loosening.
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Nicola Baldini, Professor, Director of the Research Innovation & Technology Department, Istituto Ortopedico Rizzoli
Other Study IDs: TAS-ASEPTIC
Record Dates: First submitted 2021-02-16; First posted 2021-02-26 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Loosening, Prosthesis
Keywords: Hip arthroplasty; Infection; Microbiota; Next Generation Sequencing
MeSH Terms: conditions — Prosthesis Failure; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — tissue, oral mucosa, stools
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Microbiological analysis of periprosthetic tissue — Microbiological culture of tissue samples collected intraoperatively from the newly-formed joint capsule, between prosthesis stem and femoral bone, and between the acetabular prosthesis and iliac bone.
Diagnostic Test: Histological analysis of periprosthetic tissue — Histological assessment of cellular reactivity associated with the infection on tissue samples collected intraoperatively from the newly-formed joint capsule, between prosthesis stem and femoral bone, and between the acetabular prosthesis and iliac bone.
Other: Characterization of tissue microbiota — Assessment of tissue microbiome composition using the "next-generation sequencing" of DNA extracted from samples collected intraoperatively from the newly-formed joint capsule, between prosthesis stem and femoral bone, and between the acetabular prosthesis and iliac bone.
Other: Characterization of gut microbiota — Assessment of gut microbiome composition using the "next-generation sequencing" of DNA extracted from stool samples.
Other: Characterization of oral microbiota — Assessment of oral microbiome composition using the "next-generation sequencing" of DNA extracted from a buccal swab obtained by rubbing the mucosa of cheeks, gingivae, and palate.

SUMMARY:
Recent data showed that the rate of periprosthetic infections in patients undergoing a hip arthroplasty revision for aseptic loosening is higher than what can be ascertained with conventional methods.

The study aims to assess the adequacy of next-generation sequencing of 16s ribosomal ribonucleic acid (rRNA) gene amplicons for identifying occult infections and improving the diagnostic workup. Moreover, additional testing has been planned in order to increase knowledge on the etiopathogenesis of infection.

DETAILED DESCRIPTION:
Periprosthetic infection following hip arthroplasty is one of the main causes of implant failure that leads to multiple surgical interventions, prolonged hospitalization, and higher complication rate and mortality.

Recent data prove that the rate of periprosthetic infections is higher than what can be ascertained with conventional techniques and highlight as analytical methods that allow an early and accurate diagnosis may help clinicians identify effective treatment and mitigate the devastating consequences.

New technologies based on culture-independent assays, i.e., the next-generation sequencing (NGS) of 16s rRNA gene amplicons, have entered medical microbiology as an alternative to traditional bacterial identification methods. NGS has been proven to detect microorganisms in culture-negative periprosthetic joint infection and seems to be a valid adjunct in identifying causative pathogens in samples from patients undergoing a hip arthroplasty revision for aseptic loosening.

The microbiota profiling using NGS may also help identify patients prone to develop infections. In predisposing clinical conditions, i.e., obesity and diabetes, the metabolic and nutritional alterations modify the composition and the immunomodulatory properties of intestinal microbiota. Saprophytic, non-pathogenic microorganisms usually found in the intestine and oral cavity can be transferred to other areas becoming a potential source of periprosthetic infection.

Additionally, microorganisms may live in the periprosthetic microenvironment without giving signs of overt infection. However, bacterial products, i.e., "microbe-associated molecular patterns" (MAMPs) or "pathogen-associated molecular patterns "(PAMPs), adhere to the implant surface or the wear particles and may elicit a local inflammatory response characterized by the presence of cells capable of producing cytokines that promote osteoclastogenesis, periprosthetic resorption and consequent loosening of the implant.

In summary, the current knowledge suggests that the hip arthroplasty loosening, classified as aseptic according to the preoperative clinical and laboratory investigations, could be directly or indirectly associated with infectious pathogenesis even if the microbial cultures on periprosthetic tissues are negative.

The investigators designed a small-scale study to assess the adequacy of NGS for identifying occult infections and improving the diagnostic workup in patients undergoing a hip arthroplasty revision for aseptic loosening. Moreover, additional testing has been planned to enhance knowledge on the role of unusual or difficult-to-cultivate microorganisms in the etiopathogenesis of implant failure.

ELIGIBILITY:
Inclusion Criteria:

Hip arthroplasty revision for aseptic loosening, diagnosis determined as probable according to the following criteria:

* pain and/or functional impairment;
* radiographic signs of osteolysis following wear of the implant components, or cortical reaction, or periprosthetic bone resorption;
* negative evaluation by the infectious disease specialist.

Exclusion Criteria:

* presence of a sinus tract communicating with the arthroplasty;
* bacteria isolation from aspirates or blood cultures performed preoperatively;
* serum C-reactive protein higher than 10 mg/L;
* recurrent implant dislocations;
* prosthetic fracture;
* medical history for septic arthritis, osteomyelitis;
* infections in anatomic areas other than hip;
* antibiotic therapy in the 15 days prior to surgery (with the exception of preoperative antibiotic prophylaxis);
* chronic treatment with immunosuppressive drugs;
* medical contraindications for executing sample collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients admitted at the 1st Orthopaedic and Traumatology Unit of the Istituto Ortopedico Rizzoli (Bologna, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Identification of microorganisms by microbiological cultures (number of patients with positive microbiological culture). | Within two week of admission
  Tissue samples will be sent for microbiological cultures and treated for the isolation of aerobic and anaerobic pathogens. The existence of two positive cultures will be considered to be diagnostic for periprosthetic infection; a single positive culture may occur from a contaminating organism and will be considered in conjunction with other markers of infection, including histological features.
Number of patients with histological features of periprosthetic infection | Within two week of admission
  The presence of a periprosthetic infection will be established according to the number of polymorphonuclear cells (PMN) counted in ten high-power fields (HPF) (400 × magnification, field diameter 0.54 mm)- Uninfected: 0-5 PMNs in 10 HPFs; borderline, but probably not infected: 6-10 PMNs for 10 HPF; borderline, but probably infected: >10 PMNs for 10 HPFs (but not > 5 PMNs in a single HPF); infected > 5 for HPF.
Identification of microorganisms by next-generation sequencing (NGS) (number of patients with positive NGS). | Through study completion, an average of 6 months.
  The NGS will be employed to characterize the overall microbiome profile in tissue samples, and bioinformatics used to determine the taxonomic and phylogenetic affiliation, alpha-diversity (ecological diversity of a single sample according to the number of different taxa and their relative abundances), and beta-diversity (differences in microbial community composition between samples).

SECONDARY OUTCOMES:
Characterization of taxonomic and phylogenetic affiliation of gut microbiota | Through study completion, an average of 6 months.
  The NGS technology will be employed to characterize the overall microbiome profile in stool samples, and bioinformatics used to determine the taxonomic and phylogenetic affiliation.
Characterization of alpha-diversity and beta-diversity of gut microbiota | Through study completion, an average of 6 months.
  The NGS technology will be employed to characterize the overall microbiome profile in stool samples, and bioinformatics used to determine alpha-diversity (ecological diversity of a single sample according to the number of different taxa and their relative abundances) and beta-diversity (differences in microbial community composition between samples).
Characterization of taxonomic and phylogenetic affiliation of oral microbiota | Through study completion, an average of 6 months.
  The NGS technology will be employed to characterize the overall microbiome profile in oral swab, and bioinformatics used to determine the taxonomic and phylogenetic affiliation.
Characterization of alpha-diversity and beta-diversity of oral microbiota | Through study completion, an average of 6 months.
  The NGS technology will be employed to characterize the overall microbiome profile in oral swab, and bioinformatics used to determine alpha-diversity (ecological diversity of a single sample according to the number of different taxa and their relative abundances) and beta-diversity (differences in microbial community composition between samples
Number of patients with inflammatory cellular reactivity related to bacterial products. | Through study completion, an average of 6 months.
  The inflammatory cellular reactivity proved by the presence of activated macrophages and Toll-like-receptor positive cells.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Baldini, Principal Investigator — University of Bologna, Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Background] Goswami K, Parvizi J. Culture-negative periprosthetic joint infection: is there a diagnostic role for next-generation sequencing? Expert Rev Mol Diagn. 2020 Mar;20(3):269-272. doi: 10.1080/14737159.2020.1707080. Epub 2019 Dec 24. No abstract available. PMID 31858850
- [Background] Tarabichi M, Shohat N, Goswami K, Alvand A, Silibovsky R, Belden K, Parvizi J. Diagnosis of Periprosthetic Joint Infection: The Potential of Next-Generation Sequencing. J Bone Joint Surg Am. 2018 Jan 17;100(2):147-154. doi: 10.2106/JBJS.17.00434. PMID 29342065
- [Background] Pajarinen J, Jamsen E, Konttinen YT, Goodman SB. Innate immune reactions in septic and aseptic osteolysis around hip implants. J Long Term Eff Med Implants. 2014;24(4):283-96. doi: 10.1615/jlongtermeffmedimplants.2014010564. PMID 25747031